CLINICAL TRIAL: NCT05911919
Title: Validation of a Prognostic Biomarker Using Brain Diffusion MRI in X-linked Adrenoleukodystrophy
Acronym: CALDIFF
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Braintale (Industry)
Responsible Party: Sponsor
Other Study IDs: APHP220801; IDRCB (Other: 2022-A02265-38)
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: X-linked Adrenoleukodystrophy
Keywords: Cerebral adrenoleukodystrophy (CALD); adrenomyeloneuropathy (AMN); ABCD1; MRI; Diffusion Tensor Imaging (DTI); Brain-Quant; Male; Adult
MeSH Terms: conditions — Adrenoleukodystrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Only for Patient group : Plasma and PBMC (Peripheral Blood Mononuclear Cells) collections
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients with ABCD1 pathogenic variant
  Interventions: Device: brainQuant module of brainTale-care platform
- Healthy volunteers: Healthy volunteers inclusion in order to calibrate the MRI machine used and its settings.

INTERVENTIONS:
Device: brainQuant module of brainTale-care platform — brainQuant is a software module of brainTale-care medical device (a medical device software as a service (web platform) ) for the automatic processing of brain diffusion Magnetic resonance images and the provision of the diffusion regional standardised parameters.
  Groups: Patients

SUMMARY:
CALD is an inflammatory demyelinating disease that causes severe motor and cognitive deficit leading to rapid death. Hematopoietic stem cell transplantation (HSCT) can halt neuroinflammation in CALD through the replacement of microglia (i.e., brain immune system) but only if performed during its early phase.

Using standard brain MRI, it is estimated that only 30% of adult CALD patients are identified. Complex and lengthy clinical evaluations together with MRI reading from experts improve CALD detection but are not available in routine clinical practice.

Diffusion tensor imaging is a quantitative microstructural technique that can identify neuroinflammation at a very early stage. Still, its implementation in clinical practice has been very limited due to high inter-center measurements variability and bias due to data quality issues. The approach we will use solves these problems by introducing an automatic calibration and standardization with systematic quality control enabling the use of all MRI scanners in clinical settings.

The innovative aspect of this project lies on the validation of an expert-independent prognosis biomarker able to specifically identify patients at high-risk to convert to CALD so that treatment can be initiated at the early stage of neuroinflammation.

We aim to demonstrate that this tool has at least a 2-fold sensitivity compared to the current standard of care.

DETAILED DESCRIPTION:
X-linked adrenoleukodystrophy (ALD, ORPHA:43, prevalence 1/15,000) is a rare white matter degenerative disease caused by pathogenic variants in the ABCD1 gene localised on the X chromosome. All men carrying ABCD1 pathogenic variants develop a slowly progressive myeloneuropathy (adrenomyeloneuropathy, AMN) in adulthood. Furthermore, men carrying ABCD1 pathogenic variants may also present with a rapidly progressive inflammatory leukodystrophy called cerebral ALD (CALD). Because ABCD1 variants do not predict the risk of CALD, the current standard of care is to annually monitor disease evolution by performing brain MRI and clinical evaluation to detect CALD conversion.

In adults, the inconsistency of Gadolinium contrast enhancement - the main CALD diagnosis criterion - and the presence of diffuse increase in signal of the white matter related to AMN, make the detection of true inflammatory hypersignals of the white matter (scored with the Loes score) increasingly difficult, and subject to inter-observer and inter-machine variability. Due to these limitations, and since standard MRI does not quantify myelin content or axonal injury, expert centres complement their imaging data with a battery of clinical tests - i.e., Adult ALD Clinical Scale (AACS) and Expanded Disability Severity Score (EDSS) - and neuropsychological testing to determine the disease stage of each patient with the aim to propose the best therapeutic options.

When CALD is not treated, inflammatory demyelinating lesions will cause severe motor and cognitive deficit and patients bear the risks to die within 2 to 3 years. The medical procedure of choice for males with CALD is allogenic hematopoietic stem cell transplantation (AlloHSCT) as it can stop the progression of demyelinating lesions, but only if performed during the early phase of the disease, when patients have minimal brain lesions and no or minor clinical symptoms. This treatment is ineffective or even harmful in patients in advanced stages due to the toxicity related to myeloablation protocols. In the current standard of care, the lack of early diagnostic biomarkers of CALD hampers the optimal use of AlloHSCT resulting in almost 50% mortality in adults developing CALD.

Thus, there is a crucial need for novel sensitive techniques or biomarkers easily deployable in clinical routine allowing to identify as early as possible the acute demyelinating process underlying CALD conversion.

This study aims to validate the use of an imaging biomarker, RD-index19-change, as an early diagnostic biomarker for CALD. This marker is an integrated measure of changes in cerebral regional radial diffusivity (RD) calculated from Diffusion Tensor Imaging (DTI). The RD-index19-change biomarker available in brainTale-care, a medical device developed by brainTale, can be automatically computed from MRI acquisition data in clinical routine.

The study aims to demonstrate that RD-index19-change of at least 1 point between two consecutive annual measurements has a sensitivity significantly greater than 60% and specificity significantly greater than 80%, as Objective Performance Criteria, to detect CALD conversion before or at the same time as the best experts in the field of CALD diagnosis.

The reference diagnosis of CALD will be established by an expert committee comprising 3 experts in neuroradiology, white matter diseases and CALD, based on the following information:

* One-year progression of white matter brain lesions as quantified by a Loes score change and/or the appearance of Gadolinium enhancement. The Loes scoring will be performed by an expert neuroradiologist trained to identify specific ALD lesion changes. Experts will have access to FLAIR and T1 pre- and post-contrast images.
* Increase of AACS, and especially the cerebral domain of AACS, C-AACS.
* The general disability scale EDSS
* Neuropsychological tests to evaluate processing speed, recall memory, anxiety (State-Trait Anxiety Inventory) and depression (Beck Depression Inventory)

In order for the reference diagnosis to be independent of the biomarker results, the expert committee will be blinded to the results of RD-index19-change.

The experts will also be blinded to the results of other potential biomarkers of CALD conversion that will be evaluated as secondary endpoints, i.e., plasma NfL and other DTI biomarkers (FA-index19-change, MD-index19-change and AD-index19-change).

RD-index19_change from yearly visit to yearly visit will be automatically computed from DTI acquisitions. It will therefore be independent from any clinical information or expert assessment.

The confirmation by this study that RD-index19-change can reliably detect CALD at an early stage of cerebral demyelination in an expert-independent manner will allow that:

* More CALD patients can be detected early enough to undergo AlloHSCT. The RD-index19-change should at least double the number of patients efficiently treated for this devastating neurodegenerative condition.
* Thanks to the early detection using the RD-index19-change, patients will face a decreased risk of morbidity and mortality due to AlloHSCT itself
* Patients can be followed wherever they live in France as the acquisition of MRI data for RD-index19-change calculation can be achieved on every local MR scanner after simple initial calibration.
* Besides the validation of the RD-index19-change, the CALDIFF study will greatly increase the awareness of patients, but also neurologists, about the risk of CALD in ABCD1-mutated men on a nationwide scale

ELIGIBILITY:
Patients:

Inclusion criteria

* > 18 years old
* Male gender
* Genetically diagnosed with ALD by carrying an ABCD1 pathogenic variant
* Signed written informed consent
* Affiliation to a social security regime (patient with AME cannot be included)

Exclusion criteria

* Patient with non-arrested CALD
* Other neurological conditions such as brain tumour, stroke or a traumatic head injury
* Contraindication to MRI (claustrophobia, implanted metal components in the head, panic disorder, epilepsy)
* People under legal protection measure (tutorship, curatorship or safeguard measures)
* Patient included in another interventional clinical trial

Healthy volunteers

Inclusion criteria

* Male or female subject from 18 to 65 years old
* In general good health condition
* Signed written informed consent
* Affiliation to a social security regime (healthy volunteers with AME cannot be enrolled)

Exclusion criteria

* People under legal protection measure (tutorship, curatorship or safeguard measures)
* Contraindication to MRI (claustrophobia, implanted metal components in the head, panic disorder, epilepsy)
* History of previous brain disease (including but not limited to cranial trauma in the last 12 months, glioma, stroke, neurodegenerative diseases)
* Arterial hypertension as defined in WHO criteria
* Volunteer included in another interventional clinical trial
* Pregnancy and breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients: Adult males carrying an ABCD1 pathogenic variant. Since ABCD1 is localised in X chromosome, CALD affects quasi-exclusively the male population and less than 1% of ABCD1 female carriers are at risk to develop the cerebral inflammatory form of the disease
Study Population: Adult males carrying an ABCD1 pathogenic variant
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of RD-index19 change of at least 1 point between two consecutive annual measurements to diagnose CALD before or at the same time than the reference diagnostic made by an expert committee | 1 year, 2 years, 3 years
  The expert committee comprising 3 experts in neuroradiology blinded to the RD-index19 change results.
  The study aims to demonstrate that RD-index19-change of at least 1 point between two consecutive annual measurements has a sensitivity significantly greater than 60% to detect CALD conversion before or at the same time as the best experts in the field of CALD diagnosis.
Specificity of RD-index19 change of at least 1 point between two consecutive annual measurements with repect to CALD conversion before or at the same time than the reference diagnostic made by an expert committee | 1 year, 2 years, 3 years
  The expert committee comprising 3 experts in neuroradiology blinded to the RD-index19 change results.
  The study aims to demonstrate that RD-index19-change of at least 1 point between two consecutive annual measurements has a specificity significantly greater than 80% with repect to CALD conversion before or at the same time as the best experts in the field of CALD diagnosis.

SECONDARY OUTCOMES:
Sensitivity values of plasma NfL with regard to CALD diagnosis | 1 year, 2 years, 3 years
Specificity values of plasma NfL with regard to CALD diagnosis | 1 year, 2 years, 3 years
Sensitivity values of FA-index19-change with regard to CALD diagnosis | 1 year, 2 years, 3 years
Specificity values of FA-index19-change with regard to CALD diagnosis | 1 year, 2 years, 3 years
Sensitivity values of MD-index19-change with regard to CALD diagnosis | 1 year, 2 years, 3 years
Specificity values of MD-index19-change with regard to CALD diagnosis | 1 year, 2 years, 3 years
Sensitivity values of AD-index19-change with regard to CALD diagnosis | 1 year, 2 years, 3 years
Specificity values of AD-index19-change with regard to CALD diagnosis | 1 year, 2 years, 3 years
Correlation between the clinical markers of reference in ALD (AACS (Adult ALD Clinical Scale) and EDSS (Expanded Disability Status Scale)) and RD-index19-change | 1 year, 2 years, 3 years
Correlation between the clinical markers of reference in ALD (AACS and EDSS) and FA-index19-change | 1 year, 2 years, 3 years
Correlation between the clinical markers of reference in ALD (AACS and EDSS) and MD-index19-change | 1 year, 2 years, 3 years
Correlation between the clinical markers of reference in ALD (AACS and EDSS) and AD-index19-change | 1 year, 2 years, 3 years
Correlation between the Loes score (i.e., imaging marker of reference in ALD) and RD-index19-change | 1 year, 2 years, 3 years
Correlation between the Loes score (i.e., imaging marker of reference in ALD) and FA-index19-change | 1 year, 2 years, 3 years
Correlation between the Loes score (i.e., imaging marker of reference in ALD) and MD-index19-change | 1 year, 2 years, 3 years
Correlation between the Loes score (i.e., imaging marker of reference in ALD) and AD-index19-change | 1 year, 2 years, 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Fanny MOCHEL, MD, PhD, Principal Investigator — APHP - Pitié-Salpêtrière Hospital

IPD SHARING:
Plan to Share IPD: Yes
The procedures enforced by the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not allow the transmission of the database, nor the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor.
Access Criteria: Researchers who provide a methodologically sound proposal.